CLINICAL TRIAL: NCT01936428
Title: Prospective Study of the Perception of Palliative Care by Relatives of Patients Treated in Oncology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2012.743
Record Dates: First submitted 2013-08-27; First posted 2013-09-06 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Palliative Care Perception
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- interview (Other)
  Interventions: Other: interview

INTERVENTIONS:
Other: interview

SUMMARY:
The purpose of this study is to evaluate (thanks to analysed interview) the perception of palliative care by relatives of patients treated in oncology.

ELIGIBILITY:
Inclusion Criteria:

* man or woman of age who is a relative of a patient treated in oncology
* subject who signed the informed consent
* subject without any legal protection measure and having health coverage

Exclusion Criteria:

* Relatives of patients already followed in the palliative care departement
* Subjects with cognitive impairment or expression;
* Not french spoken subjects
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Perception of palliative care evaluated by an interview with the investigator | 1 day
  The interview takes place the same day the subject signs the informed consent ; it lasts around 1 hour

SECONDARY OUTCOMES:
analysis of main elements to be used in the early information to patients and their families about palliative care. | 1 day